CLINICAL TRIAL: NCT04024956
Title: Prospective, Multicenter Study to Evaluate the Safety and Performance of a syntHetic Tissue Sealant in Reducing fluId lEakage Following Elective hepatobiLiary anD Pancreatic Surgery
Brief Title: Safety and Performance of a Synthetic Tissue Sealant in Reducing Fluid Leakage in Hepatobiliary and Pancreatic Surgery
Acronym: SHIELDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyganics BV (Industry)
Collaborators: Genae (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-3
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pancreatectomy; Hepatic Resection
Keywords: Hepatic resection; Distal pancreatectomy; Sealant

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, multicenter study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sealing Device (Experimental): Sealing Device applied in hepatic resection or distal pancreatectomy
  Interventions: Device: Sealing Device

INTERVENTIONS:
Device: Sealing Device — The Sealing Device is indicated for use in hepato-pancreato-biliary (HPB) surgery to reduce leakage of fluids from the site of surgery into the abdominal cavity and as an adjunctive hemostatic device to control minimal to moderate bleeding at the surgical site.

SUMMARY:
Polyganics BV (Groningen, The Netherlands), in close collaboration with University Hospital-Eppendorf (UKE) Hamburg, has developed the Sealing Device for use in hepato-pancreato-bilary (HPB) surgery to reduce leakage of fluids from the site of surgery into the abdominal cavity and as an adjunctive hemostatic device to control minimal to moderate bleeding at the surgical site. The Sealing Device has been challenged in pre-clinical testing (laboratory and in-vivo work), but has not been evaluated for safety and performance in humans.

This investigation will be conducted to clinically assess the safety and performance of Sealing Device as a means to reduce bile and pancreatic juice leakage in hepato-pancreato-bilary (HPB) surgery. Secondarily, the control of minimal to moderate bleeding will be assessed. To achieve adequate representation of the primary objective, the study will contain two separate surgical patient groups: Liver and Pancreas.

The primary objective of the study is to demonstrate safety and performance in reducing intra- and post-operative leakage (bile and pancreatic juices) by using the Sealing Device in patients undergoing elective hepatic resection or distal pancreatectomy.

The study will be conducted as an open-label, single-arm, multicenter study with a 16 months follow up. Up to 80 patients (40 liver and 40 pancreas patients) will be enrolled at up to 7 sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

Preoperative inclusion criteria:

Subjects will be eligible according the following criteria:

1. Subjects who are able to provide a written informed consent prior to participating in the clinical investigation.
2. Subjects who are ≥ 18 years old.
3. Subjects who are able to comply with the follow-up or other requirements.
4. Subjects who are planned for an elective hepatic resection or distal pancreatectomy.

During the surgery, the patients also need to comply with the intraoperative criteria.

Intraoperative inclusion criteria:

Subjects will be eligible according the following criteria:

1. Patch is applied manually (during open procedure, conversion procedure, or laparoscopic assisted procedure).

Exclusion Criteria:

Preoperative exclusion criteria

Subjects who meet any of the following criteria will be excluded from participation:

1. Female subjects who are pregnant and/or breastfeeding.
2. Subjects with a known allergy to any of the components of the Sealing Device (Polyurethane (SDPU), 8-ArmPEG40k-SC (SDA), Disodium Hydrogen Phosphate (Na2HPO4) (BS) and DC-Green #6 (SDD)).
3. Subject with bleeding disorders requiring anti-coagulation medication (except acetylsalicylic acid).
4. Subjects who receive double-coagulation.
5. Subjects who receive peritoneal dialysis.
6. Subjects who previously required liver transplantation.
7. Subjects with a presence of systemic infection.
8. Subject who previously participated in this study, or in any investigational drug- or device study within 30 days of screening.
9. Subjects undergoing a procedure requiring an anastomosis (e.g. Klatskin tumours or Whipple).

Intraoperative exclusion criteria:

Subjects who meet any of the following criteria will be excluded from participation:

1. Subjects with multivisceral resections, except resection of spleen.
2. Not able to apply the patch(es) according to the Instructions For Use.
3. Total surgery requiring > 3 HPB Sealing Devices of 10 x 5 cm (which equals a resection surface of more than 88cm2).

   Additional for liver group:
4. Subjects with a Grade 3 or 4 of bleeding after primary closure after liver transection (Lewis 2016).
5. Subjects with liver cirrhosis Grade C on the Child-Turcotte-Pugh score.

   Additional for pancreas group:
6. Subjects with a margin of < 1 cm between the defect and the portal vein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Bile leakage | 30 days
  Incidence of post-operative bile leakage (International Study Group of Liver Surgery Bile leakage Grading Scale); categories in order of ascending severity: biochemical leak, Grade B or Grade C
Pancreatic leakage | 30 days
  Incidence of post-operative pancreatic juice leakage (International Study Group of Pancreas Surgery Grading Scale); categories in order of ascending severity: biochemical leak, Grade B or Grade C

SECONDARY OUTCOMES:
Bleeding | Day 1
  Intra-operative control bleeding
Leak-associated comorbidities | 16 months
  Incidence of leak-associated comorbidities
re-intervention | 16 months
  Incidence of re-intervention
Ease of Use | Day 1
  Ease of Use of the device as measured by questionnaire
Post-operative bile leakage | 90 and 180 days
  Incidence of post-operative bile leakage (liver only)
Post-hepatectomy haemorrhage (PHH) | 30 days
  Incidence of post-operative bleeding (liver only)
Post-operative pancreatic juice leakage | 90 and 180 days
  Incidence of post-operative pancreatic juice leakage (pancreas only)
Post-pancreatectomy haemorrhage (PPH) | 30 days
  Incidence of post-operative bleeding (pancreas only)
(Serious) Adverse Device Effects | 16 months
  Incidence of (Serious) Adverse Device Effects
Incidence of transfusion | 16 months
  Incidence of transfusion
Length of hospital stay | 30 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitats Klinikum Hamburg-Eppendorf, Hamburg
  - University Hospital Oldenburg, Oldenburg

IPD SHARING:
Plan to Share IPD: No